CLINICAL TRIAL: NCT06508073
Title: Neural Therapy in Notalgia Paresthetica
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 4446
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Notalgia Paresthetica
Keywords: back pain; intralesional injection; neuralgia; pruritus
MeSH Terms: conditions — Back Pain; Neuralgia; Pruritus | interventions — Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neural Therapy — The injection was prepared using a solution of lidocaine 2% and saline 0.9%. A 0.4% lidocaine solution was prepared by diluting 1 cc of lidocaine with 4 cc of saline.

SUMMARY:
Patients diagnosed with Notalgia paresthetica and who received neural therapy within the last year were retrospectively screened. In the evaluations before treatment and at the 3rd month after treatment; Numerical rating scale for pain, PainDETECT questionnaire for neuropathic pain, SF-12 for quality of life and 5-D itch scale for itch level were used.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a hyperpigmented skin lesion consistent with NP
* minimum 6 months for duration of disease
* 30-60 aged
* application of neural therapy in a manner appropriate to the diagnosis

Exclusion Criteria:

* history of previous surgery or injection in the thoracic region
* presence of another treatment in the same period
* presence of any cardiac or pulmonary disease, malignancy, or advanced psychiatric disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30-60 years old patients with Notalgia Paresthetica
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale for Pain | 12 weeks after treatment
  A scale between 0 and 10 was used to question the pain level.
PainDETECT Questionnaire for assessing Neuropathic pain | 12 weeks after treatment
  The questionnaire consists of 9 items and is completed by the patient (no clinical examination is required)[1][3]. There are 7 weighted sensory descriptor items (never to very strongly) and 2 items relating to spatial and temporal pain characteristics[3]. A total score of 19 or more is indicative of likely neuropathic pain.
Short Form-12 for Quality of life | 12 weeks after treatment
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
5-D Itch Scale | 12 weeks after treatment
  The 5-D itch scale is a 5-domain disease-specific instrument evaluating the duration, degree (severity), direction (improving, unaltered or worsening), disability (impact on sleep, leisure/social, housework/errands and school/work activities) and distribution (body part affected)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)